CLINICAL TRIAL: NCT06469567
Title: Doctor's Counselling Using Culturally-responsive Pamphlet Increased Mammogram Uptake Among Malay-Muslim Women in Singapore: A Randomized Controlled Trial in a Primary Healthcare Clinic
Brief Title: Doctor's Counselling Using Culturally-responsive Pamphlet Increased Mammogram Uptake Among Malay-Muslim Women in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Polyclinics, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2020/01244
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The target group received "enhanced intervention" in the form of culturally appropriate pamphlets/flipchart and doctor counselling.
  Interventions: Other: Patient Counselling
- Control Arm (Placebo Comparator): The control group will receive the usual standard of care without the enhanced intervention.
  Interventions: Other: Patient Counselling

INTERVENTIONS:
Other: Patient Counselling — Doctor's counselling using Culturally-responsive pamphlet

SUMMARY:
Investigators conducted a randomized controlled trial to evaluate effectiveness of doctor's counselling using a culturally-responsive pamphlet in increasing mammogram uptake among Malay-Muslim women attending the clinic. Those in intervention arm received 8-minutes doctor's counselling on mammogram and breast cancer while those in control arm received 8-minutes doctor's counselling on usual care - dietary care. Investigators recruited 319 Malay-Muslim women aged 50-69 years old who have not undergone a mammogram in the past 2 years. Investigators used Poisson regression to determine effectiveness of intervention in increasing mammogram uptake and to determine any change in knowledge, perceptions and faith-based beliefs on breast cancer and mammogram after counselling.

DETAILED DESCRIPTION:
A randomized control trial was conducted at Jurong Polyclinic with the intervention arm receiving the enhanced culturally appropriate intervention, and the control arm, the usual standard of care for mammography.

Inclusion criteria Malay-Muslim women aged 50-69 years who are citizens and permanent residents of Singapore without known history of breast cancer and have not undergone screening in the last two years will be eligible for the study. These participants were recruited from Jurong Polyclinic when they came for their chronic or acute care needs.

A written informed consent was taken.

Intervention:

The target group received "enhanced intervention" in the form of culturally appropriate pamphlets/flipchart (Annex 1) and doctor counselling. After the counselling, all the women in the intervention group were referred to the staff-in-charge for a mammogram appointment in the polyclinic where they will be able to make an appointment voluntarily. All appointments were given within a period of 3 to 4 weeks. They were also given a pamphlet on breast cancer and mammogram as reinforcement after the counselling.

The control group received the usual standard of care without the "enhanced intervention".

However, they received a "placebo-attention" based on the "Healthy eating guide". Patients in this group took their own initiative to make an appointment for a mammogram.

The counselling to both groups was of a similar duration to control for Hawthorne effect.

Data collection:

Enrolment of eligible participants was by successive presentation at the polyclinic. Single blinding of the participants was done.

Anonymity was maintained by issuing unique identification numbers to all subjects.

Data was collected at baseline and 6 to 8 weeks after intervention. This interval duration is due to limitation of the time frame of the study for the practicum.

The participants filled out a self-administered questionnaire available in Malay, at baseline, to assess their knowledge, attitude, misinformation and perceptions about mammogram. Assistance was given when there was any lack of understanding.

Both the intervention and control groups were advised to come to the polyclinic for follow-up at 6 to 8 weeks. The same self-administered questionnaire on their knowledge, attitude, misinformation and perceptions about mammogram and breast cancer was given to the participants for completion. They were also asked on whether they have gone for a mammogram in the last 6-8 weeks post-intervention. This self-reported mammogram was validated with the medicals records of having had a mammogram.

When the post intervention follow-up at the polyclinic is not possible, an outreach via phone call was done to collect data.

Steps were taken to minimize social desirability bias.

ELIGIBILITY:
Inclusion Criteria:

* Malay-Muslim women aged 50-69 years
* Citizens and permanent residents of Singapore without known history of breast cancer and have not undergone screening in the last two years

Exclusion Criteria:

* All those except Malay-Muslim women aged 50-69 years who are citizens and permanent residents of Singapore without known history of breast cancer and have not undergone screening in the last two years.
* Pregnant women

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 319 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Number of participants who did a mammogram after imparting intervention. | within 6 weeks of enrolment and intervention(both done on the same day
  The mammogram uptake was assessed from patient input and verified by Radiographer

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Lather, Principal Investigator — National University Polyclinics (NUP)
Locations (1):
- National University Polyclinics, Singapore, Singapore